CLINICAL TRIAL: NCT02247531
Title: A Phase III, Multicenter, Randomized, Double-Masked, Sham-Controlled Study to Assess the Efficacy and Safety of Lampalizumab Administered Intravitreally to Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: A Study Investigating the Safety and Efficacy of Lampalizumab Intravitreal Injections in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Acronym: SPECTRI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GX29185; 2014-000106-35 (EudraCT Number)
Record Dates: First submitted 2014-07-15; First posted 2014-09-25 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — lampalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Lampalizumab once in every 4 weeks (Q4W) (Experimental): Participants will receive 10 mg (milligrams) dose of lampalizumab by intravitreal injection, Q4W, starting at the Day 1 visit for approximately 92 weeks.
  Interventions: Drug: Lampalizumab
- Lampalizumab once in every 6 weeks (Q6W) (Experimental): Participants will receive 10 mg dose of lampalizumab by intravitreal injection, Q6W, starting at the Day 1 visit for approximately 90 weeks.
  Interventions: Drug: Lampalizumab
- Sham Comparator (Sham Comparator): Participants will receive sham comparator, Q4W, starting at the Day 1 visit for approximately 92 weeks or Q6W, starting at the Day 1 visit for approximately 90 weeks.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: Lampalizumab — 10 mg dose of lampalizumab administered intravitreally.
  Other Names: RO5490249
  Arms: Lampalizumab once in every 4 weeks (Q4W); Lampalizumab once in every 6 weeks (Q6W)
Other: Sham Comparator — A sham injection is a procedure that mimics an intravitreal injection of lampalizumab.
  Arms: Sham Comparator

SUMMARY:
This study is a Phase III, double-masked, multicenter, randomized, sham injection-controlled study evaluating the efficacy and safety of lampalizumab administered by intravitreal injections in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Participants aged greater than or equal to (>/=) 50 years
* Well demarcated area(s) of Geographic Atrophy (GA) secondary to Age-Related Macular Degeneration (AMD) with no evidence of prior or active choroidal neovascularization (CNV) in both eyes

Exclusion Criteria:

Ocular Exclusion Criteria (Study Eye):

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD
* Previous laser photocoagulation for CNV, diabetic macular edema, retinal vein occlusion, and proliferative diabetic retinopathy
* Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection, anti-angiogenic drugs, anti-complement agents, or device implantation)

Ocular Exclusion Criteria (Both Eyes):

* GA in either eye due to causes other than AMD
* Previous treatment with eculizumab, lampalizumab, and/or fenretinide

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 975 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (153):
- United States (67):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - UCSD Shiley Eye Center, La Jolla, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - N CA Retina Vitreous Assoc, Mountain View, California
  - Byers Eye Insitute at Stanford, Palo Alto, California
  - Retina Consultants, San Diego, Poway, California
  - University of California, Davis, Eye Center, Sacramento, California
  - Retinal Consultants Med Group, Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - University of Colorado, Aurora, Colorado
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Colorado Retina Associates, PC, Golden, Colorado
  - New England Retina Associates, Hamden, Connecticut
  - Retina Group of New England, Waterford, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Retina Health Center, Fort Myers, Florida
  - Bascom Palmer Eye Institute, Naples, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Vitreo Retinal Consultants, Wichita, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - The Retina Care Center, Baltimore, Maryland
  - Wilmer Eye Institute, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Retina Specialists, Towson, Maryland
  - Mass Eye and Ear Infirmary, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Kresge Eye Institute, Detroit, Michigan
  - Vitreoretinal Surgery, Edina, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - UNMC Truhlsen Eye Institute, Omaha, Nebraska
  - Sierra Eye Associates, Reno, Nevada
  - Mid Atlantic Retina - Wills Eye Hospital, Cherry Hill, New Jersey
  - Retinal & Ophthalmic Cons PC, Northfield, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - New York Weil Cornell Med Ctr, New York, New York
  - Vitreous-Retina-Macula, New York, New York
  - Retina Assoc of Western NY, Rochester, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Duke University Eye Center; Vitreoretinal, Durham, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - OSU Eye Physicians & Surgeons, Columbus, Ohio
  - Retina & Vitreous Center of Southern Oregon, Ashland, Oregon
  - Retina Northwest, Portland, Oregon
  - Oregon HSU; Casey Eye Institute, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Allegheny Ophthalmic & Orbital, Pittsburgh, Pennsylvania
  - MUSC Storm eye institute, Charleston, South Carolina
  - Palmetto Retina Center, Florence, South Carolina
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Charles Retina Institution, Germantown, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Scott and White Hospital, Temple, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Univ of Virginia Ophthalmology, Charlottesville, Virginia
  - Vitreoretinal Associates of Washington, Bellevue, Washington
- Argentina (3):
  - Oftalmos, Capital Federal
  - Instituto de la Vision, Capital Federal
  - Hospital El Cruce, San Juan Bautista
- Australia (5):
  - Queensland Eye Institute, Brisbane, Queensland
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Vision Eye Institute Eastern, Box Hill, Victoria
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Medizinische Universität Wien; Universitätsklinik für Augenheilkunde und Optometrie, Vienna, Austria
- Belgium (2):
  - CHU Brugmann (Victor Horta), Brussels
  - UZ Leuven Sint Rafael, Leuven
- Glostrup Hospital, Øjenafdelingen, Forskningsafsnit Ø37, Glostrup Municipality, Denmark
- France (6):
  - Hopital Pellegrin; Ophtalmologie, Bordeaux
  - CHU Bocage; Ophtalmologie, Dijon
  - Hopital de la croix rousse; Ophtalmologie, Lyon
  - Centre Paradis Monticelli; Ophtalmologie, Marseille
  - Hopital Hotel Dieu Et Hme; Clinique Ophtalmologique, Nantes
  - CHNO des Quinze Vingts; Ophtalmologie, Paris
- Germany (8):
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitätsklinik Heidelberg; Augenklinik, Heidelberg
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH; Augenklinik, Ludwigshafen
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Augenklinik und Poliklinik, Mainz
  - LMU Klinikum der Universität, Augenklinik, München
  - Klinikum rechts der Isar der TU München; Augenklinik, München
  - Universitätsklinikum Regensburg, Klinik & Poliklinik für Augenheilkunde, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (3):
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont, Szemeszet KR, Budapest
  - Semmelweis Egyetem AOK, Szemeszeti Klinika, Budapest
  - Ganglion Medial Center, Pécs
- Italy (6):
  - UNIVERSITA' DEGLI STUDI DI GENOVA - Di.N.O.G.;CLINICA OCULISTICA, Genoa, Liguria
  - Irccs Ospedale San Raffaele;U.O. Oculistica, Milan, Lombardy
  - ASST FATEBENEFRATELLI SACCO; Oculistica (Sacco), Milan, Lombardy
  - A.S.L. to1 Presidio Ospedaliero Sperino Oftalmico, Turin, Piedmont
  - Azienda Ospedaliero-Universitaria Careggi; S.O.D. Oculistica, Florence, Tuscany
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Clinica Oculistica, Udine, Veneto
- Mexico (3):
  - Hospital Nuestra Señora de La Luz, Mexico City
  - Hospital Universitario de Monterrey, Monterrey
  - Instituto Mexicano de Oftalmologia I.A.P., Querétaro
- Netherlands (2):
  - Radboud University Nijmegen Medical Centre; Ophthalmology, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Peru (3):
  - Mácula D&T, Lima
  - TG Laser Oftalmica, Lima
  - Centro de Investigacion Oftalmolaser, Lima
- Poland (4):
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Szpital Specjalistyczny nr 1; Oddzial Okulistyki, Bytom
  - Klinika Okulistyczna Jasne Błonia, Lodz
  - Uniwersytecki Szpital Kliniczny; Klinika Okulistyki, Wroclaw
- Portugal (4):
  - AIBILI - Association for Innovation and Biomedical Research on Light, Coimbra
  - Espaco Medico Coimbra, Coimbra
  - Hospital de Santa Maria; Servico de Oftalmologia, Lisbon
  - Hospital de Sao Joao; Servico de Oftalmologia, Porto
- Russia (3):
  - SAHI "Republic clinical ophthalmological hospial of Ministry of Heal of Tatarstan Republic", Kazan'
  - FSBI "Scientific Research Institute of Eye Diseases" of Russian Academy of medical Sciences, Moscow
  - St. Educ.Inst. of High Prof.Education "Samara State Medical University"; Chair of ophathalmology, Samara
- Slovakia (2):
  - FNsP F. D. Roosevelta Banska Bystrica, II.Ocna klinika SZU, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Nemocnica sv. Cyrila a Metoda Ocna klinika SZU a UNB, Bratislava
- Spain (7):
  - Instituto Oftalmologico Gomez Ulla, Santiago de Compostela, LA Coruña
  - Clinica Universitaria de Navarra; Servicio de Oftalmologia, Pamplona, Navarre
  - Hospital Perpetuo Socorro; Servicio de Oftalmología, Albacete
  - Instituto de microcirugia ocular, Barcelona
  - VISSUM Madrid Santa Hortensia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oftalmologia, Madrid
  - Hospital Universitario la Fe: Servicio de Oftalmologia, Valencia
- St Eriks Eye Hospital, Stockholm, Sweden
- Switzerland (2):
  - Inselspital Bern, Universitätsklinik für Augenheilkunde, Bern
  - Vista Klinik Binningen, Binningen
- Turkey (Türkiye) (6):
  - Hacettepe University Medical Faculty; Department of Ophthalmology, Ankara
  - Ankara University Medical Faculty; Department of Ophthalmology, Ankara
  - Ankara Baskent University Medical Faculty; Department of Ophthalmology, Ankara
  - Istanbul University Istanbul Medical Faculty; Department of Ophthalmology, Istanbul
  - Ege University Medical Faculty; Department of Ophthalmology, Izmir
  - Dokuz Eylul University Medical Faculty; Department of Ophthalmology, Izmir
- United Kingdom (14):
  - Royal Victoria Hospital, Belfast
  - Bradford Royal Infirmary, Bradford
  - Bristol Eye Hospital, Bristol
  - University Hospital of Wales, Cardiff
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Royal Liverpool University Hospital; St Paul's Clinical Eye Research Centre, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Kings College Hospital, London
  - Macular Treatment Centre; Royal Eye Hospital, Manchester
  - Hillingdon Hospital, Middx
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Southampton General Hospital, Southampton
  - The Royal Wolverhampton Hospitals NHS Trust, Wolverhampton
  - The York Hospital, York

REFERENCES:
- [Derived] Salvi A, Cluceru J, Gao SS, Rabe C, Schiffman C, Yang Q, Lee AY, Keane PA, Sadda SR, Holz FG, Ferrara D, Anegondi N. Deep Learning to Predict the Future Growth of Geographic Atrophy from Fundus Autofluorescence. Ophthalmol Sci. 2024 Oct 23;5(2):100635. doi: 10.1016/j.xops.2024.100635. eCollection 2025 Mar-Apr. PMID 39758130
- [Derived] Cluceru J, Anegondi N, Gao SS, Lee AY, Lad EM, Chakravarthy U, Yang Q, Steffen V, Friesenhahn M, Rabe C, Ferrara D. Topographic Clinical Insights From Deep Learning-Based Geographic Atrophy Progression Prediction. Transl Vis Sci Technol. 2024 Aug 1;13(8):6. doi: 10.1167/tvst.13.8.6. PMID 39102242
- [Derived] Bressler NM, Freund KB, Bakri SJ, Kim JE, Ferrara D, Brittain C, Pickthorn K, Lin H, Sun C, Martin J. Intraocular Pressure Outcomes After Lampalizumab Injections in Patients With Geographic Atrophy. JAMA Ophthalmol. 2024 Aug 1;142(8):772-776. doi: 10.1001/jamaophthalmol.2024.2061. PMID 38900484
- [Derived] Chang DS, Callaway NF, Steffen V, Csaky K, Guymer RH, Birch DG, Patel PJ, Ip M, Gao SS, Briggs J, Honigberg L, Lai P, Ferrara D, Sepah YJ. Macular Sensitivity Endpoints in Geographic Atrophy: Exploratory Analysis of Chroma and Spectri Clinical Trials. Ophthalmol Sci. 2023 Jun 12;4(1):100351. doi: 10.1016/j.xops.2023.100351. eCollection 2024 Jan-Feb. PMID 37869030
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- [Derived] Heier JS, Pieramici D, Chakravarthy U, Patel SS, Gupta S, Lotery A, Lad EM, Silverman D, Henry EC, Anderesi M, Tschosik EA, Gray S, Ferrara D, Guymer R; Chroma and Spectri Study Investigators. Visual Function Decline Resulting from Geographic Atrophy: Results from the Chroma and Spectri Phase 3 Trials. Ophthalmol Retina. 2020 Jul;4(7):673-688. doi: 10.1016/j.oret.2020.01.019. Epub 2020 Jan 31. PMID 32199866
- [Derived] Holz FG, Sadda SR, Busbee B, Chew EY, Mitchell P, Tufail A, Brittain C, Ferrara D, Gray S, Honigberg L, Martin J, Tong B, Ehrlich JS, Bressler NM; Chroma and Spectri Study Investigators. Efficacy and Safety of Lampalizumab for Geographic Atrophy Due to Age-Related Macular Degeneration: Chroma and Spectri Phase 3 Randomized Clinical Trials. JAMA Ophthalmol. 2018 Jun 1;136(6):666-677. doi: 10.1001/jamaophthalmol.2018.1544. PMID 29801123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 975 participants were randomized to the study at 144 study sites across 22 countries. The study was terminated early by the Sponsor due to lack of efficacy.
Pre-assignment Details: This study enrolled participants with bilateral Geographic Atrophy (GA) secondary to Age-Related Macular Degeneration (AMD) and no signs of prior or active choroidal neovascularization (CNV), age >= 50 years with a valid complement factor I (CFI)-profile biomarker result.
Groups:
- Sham Comparator: Participants received sham comparator, once every 4 weeks (Q4W) starting at the Day 1 visit or once every 6 weeks (Q6W) starting at the Day 1 visit.
- Lampalizumab Q4W: Participants received 10 mg (milligrams) dose of lampalizumab by intravitreal injection Q4W starting at the Day 1 visit.
- Lampalizumab Q6W: Participants received 10 mg dose of lampalizumab by intravitreal injection Q6W starting at the Day 1 visit.
Period: Overall Study
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Started | 321 | 330 | 324
Completed | 215 | 205 | 214
Not Completed | 106 | 125 | 110
Not completed — Adverse Event | 3 | 4 | 9
Not completed — Death | 8 | 9 | 5
Not completed — Lost to Follow-up | 1 | 8 | 3
Not completed — Non-compliance | 2 | 2 | 0
Not completed — Withdrawal by Subject | 26 | 31 | 25
Not completed — Study Terminated by Sponsor | 64 | 66 | 62
Not completed — Physician Decision | 0 | 2 | 2
Not completed — Unspecified Reason | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W | Total
Number analyzed (Participants) | 321 | 330 | 324 | 975
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (8.3) | 77.3 (7.8) | 78.7 (8.0) | 77.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 197 | 190 | 578
  Male | 130 | 133 | 134 | 397
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 16 | 37
  Not Hispanic or Latino | 298 | 310 | 297 | 905
  Not Stated | 7 | 8 | 8 | 23
  Unknown | 4 | 3 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 1 | 6
  Asian | 3 | 1 | 1 | 5
  Black or African American | 0 | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  White | 306 | 315 | 315 | 936
  Multiple | 2 | 0 | 1 | 3
  Unknown | 7 | 10 | 6 | 23
Geographic Atrophy (GA) Area, as Assessed by Fundus Autofluoresence (FAF) [Mean (Standard Deviation); unit: millimeter square (mm^2)] — At baseline the area of GA was assessed by FAF.
  millimeter square (mm^2) | 7.554 (3.983) | 8.308 (3.916) | 8.498 (4.260) | 8.123 (4.071)
Number of Absolute Scotomatous Points as Assessed by Mesopic Micrometry [Mean (Standard Deviation); unit: number of absolute scotomatous points] — Scotomatous points were the testing points on microperimetry examination that were centered on the macula and reported a lack of retinal sensitivity within the range tested. Mesopic microperimetry assessments were performed post-dilation on the study eye only, and the data was forwarded to the central reading center. Population: The microperimetry analysis population consisted of all participants who met the microperimetry eligibility criteria assessed by the reading center (participants at selected sites only; participants grouped according to treatment assigned at randomization).
  number of absolute scotomatous points
    number analyzed (Participants) | 48 | 58 | 55 | 161
    (all) | 23.2 (13.5) | 28.2 (17.3) | 27.9 (14.4) | 26.6 (15.3)
Macular Sensitivity as Assessed by Mesopic Microperimetry [Mean (Standard Deviation); unit: decibel (dB)] — Mesopic microperimetry was used to assess macular sensitivity and assessments were performed post-dilation on the study eye only, and the data was forwarded to the central reading center. Population: The microperimetry analysis population consisted of all participants who met the microperimetry eligibility criteria assessed by the reading center (participants at selected sites only; participants grouped according to treatment assigned at randomization).
  decibel (dB)
    number analyzed (Participants) | 48 | 57 | 54 | 159
    (all) | 6.5 (3.3) | 5.7 (3.8) | 5.3 (3.2) | 5.8 (3.5)
Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Study [Mean (Standard Deviation); unit: letters] — BCVA score was based on the number of letters read correctly on the ETDRS visual acuity chart assessed at a starting distance of 4 meters (m). BCVA score testing was performed prior to dilating the eyes. BCVA score ranges from 0 to 100 letters in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
  letters
    number analyzed (Participants) | 319 | 330 | 321 | 970
    (all) | 66.1 (9.8) | 66.0 (9.6) | 65.7 (9.8) | 66.0 (9.7)
Low Luminance Visual Acuity (LLVA) as Assessed by ETDRS Chart Under Low Luminance Conditions [Mean (Standard Deviation); unit: letters] — The LLVA was measured by placing a 2.0-log-unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart. The assessment was performed prior to dilating the eyes. Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
  letters
    number analyzed (Participants) | 310 | 322 | 310 | 942
    (all) | 36.8 (16.5) | 36.1 (17.5) | 35.8 (16.8) | 36.2 (16.9)
Binocular Reading Speed as Assessed by Minnesota Low-Vision Reading Test or Radner Reading Charts [Mean (Standard Deviation); unit: words per minute (wpm)] — Minnesota Low-Vision Reading (MNRead) acuity cards were continuous-text reading-acuity cards suitable for measuring reading acuity and reading speed of normal and low-vision participants. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. Reading test was stopped when reading time was longer than 20 seconds or when participant was making severe errors. Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
  words per minute (wpm)
    number analyzed (Participants) | 298 | 303 | 302 | 903
    (all) | 105.16 (56.94) | 104.38 (54.35) | 99.75 (56.56) | 103.09 (55.94)
Monocular Maximum Reading Speed as Assessed by MNRead Charts or Radner Reading Charts [Mean (Standard Deviation); unit: wpm] — MNRead acuity cards were continuous-text reading-acuity cards suitable for measuring reading acuity and reading speed of normal and low-vision participants. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. Reading test was stopped when reading time was longer than 20 seconds or when participant was making severe errors. Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
  wpm
    number analyzed (Participants) | 300 | 310 | 304 | 914
    (all) | 81.20 (57.48) | 80.38 (53.70) | 74.52 (50.11) | 78.70 (53.85)
National Eye Institute Visual Functioning Questionnaire 25-item (NEI VFQ-25) Version Composite Score [Mean (Standard Deviation); unit: score on a scale] — NEI-VFQ-25 questionnaire included 25 items based on which overall composite VFQ score and 12 subscales were derived: near activities, distance activities, general health,general vision, ocular pain, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision and peripheral vision. Response to each question converted to 0-100 score. Each subscale, total score=average of items contributing to score. For each subscale and total score, score range: 0 to 100, a higher score represents better functioning. Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
  score on a scale
    number analyzed (Participants) | 283 | 299 | 296 | 878
    (all) | 64.84 (15.80) | 62.88 (17.50) | 64.03 (17.65) | 63.90 (17.02)
NEI VFQ-25 Near Activity Subscale Score [Mean (Standard Deviation); unit: score on a scale] — NEI-VFQ-25 questionnaire included 25 items based on near activities, which are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf. Response to each question converted to 0-100 score. Subscale=average of items contributing to score. For this subscale the score range is 0 to 100, a higher score represents better functioning. Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
  score on a scale
    number analyzed (Participants) | 283 | 299 | 296 | 878
    (all) | 53.89 (19.91) | 51.68 (21.92) | 53.24 (22.07) | 52.92 (21.34)
NEI VFQ-25 Distance Activity Subscale Score [Mean (Standard Deviation); unit: scores on a scale] — NEI-VFQ-25 questionnaire included 25 items based on which distance activities was measured. Distance activities are defined as reading street signs or names on stores, and going down stairs, steps, or curbs. Response to each question converted to 0-100 score. Subscale=average of items contributing to score. For this subscale the score range is 0 to 100, a higher score represents better functioning. Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
  scores on a scale
    number analyzed (Participants) | 283 | 299 | 296 | 878
    (all) | 62.68 (21.41) | 58.57 (22.03) | 60.95 (21.55) | 60.70 (21.71)
Mean Functional Reading Independence (FRI) Index [Mean (Standard Deviation); unit: score on a scale] — The FRI was an interviewer-administered questionnaire with 7-items on functional reading activities most relevant to GA AMD participants. It has one total index score. For each FRI Index reading activity performed in the past 7 days, participants were asked about the extent to which they required vision aids, adjustments in the activity, or help from another participant. Mean FRI Index scores range from 1 to 4, with higher scores indicating greater independence. Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
  score on a scale
    number analyzed (Participants) | 278 | 296 | 293 | 867
    (all) | 2.70 (0.79) | 2.66 (0.82) | 2.64 (0.87) | 2.67 (0.83)
GA Area in Complement Factor I (CFI) Positive Participants [Mean (Standard Deviation); unit: mm^2] — For CFI profile, positive biomarker status refers to the presence (carrier) of the risk allele at CFI and at least one risk allele at complement factor H (CFH) or risk locus containing both complement component 2 and complement factor B (C2/CFB). Population: ITT population included all the participants who were randomized to the study. Reported here is the number of CFI-positive participants for whom data were collected.
  mm^2
    number analyzed (Participants) | 194 | 199 | 194 | 587
    (all) | 7.491 (4.068) | 8.183 (3.835) | 8.652 (4.250) | 8.109 (4.074)
GA Area in CFI Negative Participants [Mean (Standard Deviation); unit: mm^2] — For CFI profile, negative biomarker status refers to the absence of the risk allele at CFI and at least one risk allele at CFH or C2/CFB. Population: ITT population included all the participants who were randomized to the study. Reported here is the number of CFI-negative participants for whom data were collected.
  mm^2
    number analyzed (Participants) | 127 | 131 | 130 | 388
    (all) | 7.650 (3.862) | 8.499 (4.044) | 8.268 (4.281) | 8.144 (4.073)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Geographic Atropy (GA) Area, as Assessed by Fundus Autofluoresence (FAF) at Week 48
Description: The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of GA lesion area (worsening; disease progression).
Time Frame: Baseline, Week 48
Population: Intent-to-treat (ITT) population included all the participants who were randomized to the study. Participants analyzed in this outcome measure were those included in Mixed-effect model repeated measures (MMRM analysis).
Measure: Mean (Standard Error); unit: millimeter square (mm^2)
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 291 | 293 | 291
millimeter square (mm^2) | 1.932 (0.056) | 2.089 (0.056) | 2.019 (0.056)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline GA area, lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.0479, MMRM; Difference in Adjusted Means = 0.157, 95% CI 2-sided [0.001 to 0.313]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2739, MMRM; Difference in Adjusted Means = 0.087, 95% CI 2-sided [-0.069 to 0.243]

2. Secondary Outcome: Change From Baseline in Number of Absolute Scotomatous Points Assessed by Mesopic Microperimetry at Week 48
Description: Scotomatous points were the testing points on microperimetry examination that were centered on the macula and reported a lack of retinal sensitivity within the range tested. Mesopic microperimetry assessments were performed post-dilation on the study eye only, and the data was forwarded to the central reading center. A positive change from baseline indicates an increase in the number of absolute scotomatous points (more lack of retinal sensitivity); disease worsening. Data were collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: The microperimetry analysis population consisted of all participants who met the microperimetry eligibility criteria assessed by the reading center (participants at selected sites only; participants grouped according to treatment assigned at randomization). Participants analyzed in this outcome measure were those included in MMRM analysis.
Measure: Mean (Standard Error); unit: number of absolute scotomatous points
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 39 | 42 | 43
number of absolute scotomatous points | 5.4 (1.6) | 5.0 (1.5) | 6.7 (1.5)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline number of absolute scotomatous points, GA lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.8400, MMRM; Difference in Adjusted Means = -0.4, 95% CI 2-sided [-4.8 to 3.9]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5587, MMRM; Difference in Adjusted Means = 1.3, 95% CI 2-sided [-3.1 to 5.7]

3. Secondary Outcome: Change From Baseline in Macular Sensitivity as Assessed by Mesopic Microperimetry at Week 48
Description: Mesopic microperimetry was used to assess macular sensitivity and assessments were performed post-dilation on the study eye only, and the data was forwarded to the central reading center. A negative change from baseline indicates a decrease in the mean macular sensitivity; disease worsening. Data were collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Error); unit: decibel (dB)
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 39 | 41 | 42
decibel (dB) | -0.99 (0.36) | -0.89 (0.34) | -1.25 (0.35)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline mean macular sensitivity, GA lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.8358, MMRM; Difference in Adjusted Means = 0.10, 95% CI 2-sided [-0.88 to 1.09]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.6117, MMRM; Difference in Adjusted Means = -0.26, 95% CI 2-sided [-1.25 to 0.74]

4. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart at Week 48
Description: BCVA score was based on the number of letters read correctly on the ETDRS visual acuity chart assessed at a starting distance of 4 meters (m). A decrease in the VA score indicates a worsening in visual acuity. BCVA score testing was performed prior to dilating the eyes. The data was collected up to Week 48 instead of Week 96, due to early termination of the study. BCVA score ranges from 0 to 100 letters in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A negative change from baseline indicates a decrease in the visual acuity; disease worsening.
Time Frame: Baseline, Week 48
Population: ITT population included all the participants who were randomized to the study. Participants analyzed in this outcome measure were those included in MMRM analysis.
Measure: Mean (Standard Error); unit: letters
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 288 | 286 | 287
letters | -5.3 (0.7) | -4.6 (0.7) | -5.1 (0.7)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline BCVA, GA lesion location, biomarker status, and sex; Test type: Superiority; p = 0.4651, MMRM; Difference in Adjusted Means = 0.7, 95% CI 2-sided [-1.2 to 2.5]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.7885, MMRM; Difference in Adjusted Means = 0.3, 95% CI 2-sided [-1.6 to 2.1]

5. Secondary Outcome: Percentage of Participants With Less Than 15 Letters Loss From Baseline in BCVA Score at Week 48
Description: Loss of less than 15 letters from baseline was assessed by the ETDRS chart at a starting distance of 4 meters (m). Data were collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Week 48
Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
Measure: Number; unit: percentage of participants
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 288 | 286 | 287
percentage of participants | 87.1 | 88.2 | 86.8
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Test type: Superiority; p = 0.6892, Regression, Logistic; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; Test type: Superiority; p = 0.9104, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.6]

6. Secondary Outcome: Change From Baseline in Low Luminance Visual Acuity (LLVA) as Assessed by ETDRS Chart Under Low Luminance Conditions at Week 48
Description: The low luminance visual acuity was measured by placing a 2.0-log-unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart. The assessment was performed prior to dilating the eyes. A negative change from baseline indicates a decrease in the visual acuity; disease worsening. Data were collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: letters
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 274 | 278 | 274
letters | -2.5 (0.6) | -2.6 (0.6) | -3.6 (0.6)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline LLVA, GA lesion location, biomarker status, modified baseline BCVA ETDRS chart Snellen equivalent category, and sex; Test type: Superiority; p = 0.8931, MMRM; Difference in Adjusted Means = -0.1, 95% CI 2-sided [-1.8 to 1.5]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.1754, MMRM; Difference in Adjusted Means = -1.1, 95% CI 2-sided [-2.8 to 0.5]

7. Secondary Outcome: Percentage of Participants With Less Than 15 Letters Loss From Baseline in LLVA Score at Week 48
Description: Loss of less than 15 letters from baseline was assessed by the ETDRS chart at a starting distance of 4 m. Data were collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Week 48
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 274 | 278 | 274
percentage of participants | 90.1 [83.7 to 91.5] | 92.1 [86.4 to 93.5] | 89.6 [82.9 to 90.9]
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Test type: Superiority; p = 0.3707, Regression, Logistic; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.7 to 2.2]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; Test type: Superiority; p = 0.8382, Regression, Logistic; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.6 to 1.6]

8. Secondary Outcome: Change From Baseline in Binocular Reading Speed as Assessed by Minnesota Low-Vision Reading Test (MNRead) Charts or Radner Reading Charts at Week 48
Description: MNRead acuity cards were continuous-text reading-acuity cards suitable for measuring the reading acuity and reading speed of normal and low-vision participants. The MNRead acuity cards consisted of single, simple sentences with equal numbers of characters. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. The Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. The reading test was stopped when the reading time was longer than 20 seconds or when the participant was making severe errors. A negative change from baseline indicates a decrease in the binocular reading speed; disease worsening. Data were collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: words per minute (wpm)
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 261 | 255 | 266
words per minute (wpm) | -15.27 (2.33) | -13.92 (2.36) | -14.20 (2.31)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, baseline maximum reading speed, type of reading charts, baseline BCVA of better seeing eye, biomarker status, and sex; Test type: Superiority; p = 0.6841, MMRM; Difference in Adjusted Means = 1.35, 95% CI 2-sided [-5.16 to 7.85]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.7443, MMRM; Difference in Adjusted Means = 1.07, 95% CI 2-sided [-5.37 to 7.52]

9. Secondary Outcome: Change From Baseline in Monocular Maximum Reading Speed as Assessed by MNRead Charts or Radner Reading Charts at Week 48
Description: MNRead acuity cards were continuous-text reading-acuity cards suitable for measuring reading acuity and reading speed of normal and low-vision participants. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. Reading test was stopped when reading time was longer than 20 seconds or when participant was making severe errors. A negative change from baseline indicates a decrease in the monocular reading speed; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: wpm
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 264 | 264 | 272
wpm | -16.58 (2.30) | -16.46 (2.30) | -18.30 (2.27)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, baseline maximum reading speed, biomarker status, modified baseline BCVA, and sex; Test type: Superiority; p = 0.9713, MMRM; Difference in Adjusted Means = 0.12, 95% CI 2-sided [-6.28 to 6.52]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.5945, MMRM; Difference in Adjusted Means = -1.72, 95% CI 2-sided [-8.08 to 4.63]

10. Secondary Outcome: Change From Baseline in National Eye Institute Visual Functioning Questionnaire 25-item (NEI VFQ-25) Version Composite Score at Week 48
Description: NEI-VFQ-25 questionnaire included 25 items based on which overall composite VFQ score and 12 subscales were derived: near activities, distance activities, general health, general vision, ocular pain, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision and peripheral vision. Response to each question converted to 0-100 score. Each subscale or total score is the average of items contributing to the score. For each subscale and total score the score range is 0 to 100 with a higher score representing better functioning. A negative change from baseline indicates a decrease in the visual functioning; disease worsening. Data were collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 251 | 259 | 265
score on a scale | -2.08 (0.74) | -0.86 (0.73) | -1.05 (0.72)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, baseline score, baseline BCVA of better seeing eye, biomarker status, and sex; Test type: Superiority; p = 0.2438, MMRM; Difference in Adjusted Means = 1.22, 95% CI 2-sided [-0.83 to 3.27]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.3202, MMRM; Difference in Adjusted Means = 1.03, 95% CI 2-sided [-1.01 to 3.07]

11. Secondary Outcome: Change From Baseline in NEI VFQ-25 Near Activity Subscale Score at Week 48
Description: NEI-VFQ-25 questionnaire included 25 items based on which near activities were measured. Near activities are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf. Response to each question converted to 0-100 score. Subscale=average of items contributing to score. For this subscale the score range is 0 to 100, a higher score represents better functioning. A negative change from baseline indicates a decrease in the near visual activities; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 251 | 259 | 265
score on a scale | -4.12 (0.91) | -1.49 (0.89) | -1.93 (0.88)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0388, MMRM; Difference in Adjusted Means = 2.64, 95% CI 2-sided [0.14 to 5.14]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0833, MMRM; Difference in Adjusted Means = 2.20, 95% CI 2-sided [-0.29 to 4.68]

12. Secondary Outcome: Change From Baseline in NEI VFQ-25 Distance Activity Subscale Score at Week 48
Description: NEI-VFQ-25 questionnaire included 25 items based on which distance activities were measured. Distance activities are defined as reading street signs or names on stores, and going down stairs, steps, or curbs. Response to each question converted to 0-100 score. Subscale=average of items contributing to score. For this subscale the score range is 0 to 100, a higher score represents better functioning. A negative change from baseline indicates a decrease in the distance visual activities; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 251 | 259 | 265
score on a scale | -2.83 (1.04) | -1.80 (1.03) | -2.24 (1.01)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.4795, MMRM; Difference in Adjusted Means = 1.04, 95% CI 2-sided [-1.84 to 3.91]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.6822, MMRM; Difference in Adjusted Means = 0.60, 95% CI 2-sided [-2.26 to 3.45]

13. Secondary Outcome: Change From Baseline in Mean Functional Reading Independence (FRI) Index at Week 48
Description: The FRI was an interviewer-administered questionnaire with 7 items on functional reading activities most relevant to GA AMD participants. It has one total index score. For each FRI Index reading activity performed in the past 7 days, participants were asked about the extent to which they required vision aids, adjustments in the activity, or help from another participant. Mean FRI Index scores range from 1 to 4, with higher scores indicating greater independence. A negative change from baseline indicates a decrease in the FRI; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 248 | 257 | 260
score on a scale | -0.16 (0.04) | -0.12 (0.04) | -0.14 (0.04)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, baseline Mean FRI Index score, baseline BCVA of better seeing eye, biomarker status, and sex; Test type: Superiority; p = 0.5227, MMRM; Difference in Adjusted Means = 0.04, 95% CI 2-sided [-0.07 to 0.14]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.7475, MMRM; Difference in Adjusted Means = 0.02, 95% CI 2-sided [-0.09 to 0.13]

14. Primary Outcome: Change From Baseline in GA Area in Complement Factor I (CFI) Positive and Negative Participants at Week 48
Description: For CFI profile, positive or negative biomarker status refers to the presence (carrier) or absence of the risk allele at CFI and at least one risk allele at complement factor H (CFH) or risk locus containing both complement component 2 and complement factor B (C2/CFB).The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of GA lesion area (worsening; disease progression).
Time Frame: Baseline, Week 48
Population: ITT population included all the participants who were randomized to the study. The analysis was done specifically for CFI-positive and negative participants.
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 321 | 330 | 324
mm^2
  CFI-Positive Participants: number analyzed (Participants) | 176 | 183 | 172
  CFI-Positive Participants | 2.007 (0.074) | 2.057 (0.072) | 2.032 (0.073)
  CFI-Negative Participants: number analyzed (Participants) | 115 | 110 | 119
  CFI-Negative Participants | 1.809 (0.087) | 2.149 (0.087) | 1.991 (0.085)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; CFI Positive: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline GA area, lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.6333, MMRM; Difference in Adjusted Means = 0.049, 95% CI 2-sided [-0.153 to 0.252]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.8105, MMRM; Difference in Adjusted Means = 0.025, 95% CI 2-sided [-0.180 to 0.230]
Statistical Analysis 3: Comparison: Sham Comparator vs Lampalizumab Q4W; CFI Negative: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline GA area, lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.0063, MMRM; Difference in Adjusted Means = 0.340, 95% CI 2-sided [0.097 to 0.584]
Statistical Analysis 4: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p = 0.1359, MMRM; Difference in Adjusted Means = 0.182, 95% CI 2-sided [-0.058 to 0.422]

ADVERSE EVENTS:
Time Frame: Up to approximately 2 years
Description: Safety population included all participants who received at least one dose of study drug.
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
All-Cause Mortality (participants affected / at risk) | 9/318 | 10/329 | 7/323
Serious Adverse Events (participants affected / at risk) | 99/318 | 113/329 | 111/323
Other Adverse Events (participants affected / at risk) | 227/318 | 268/329 | 253/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Comparator (N=318) | Lampalizumab Q4W (N=329) | Lampalizumab Q6W (N=323)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 3
Angina unstable (Cardiac disorders) | 1 | 0 | 2
Aortic valve stenosis (Cardiac disorders) | 2 | 0 | 0
Arrhythmia (Cardiac disorders) | 2 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 7 | 2
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Atrioventricular dissociation (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 2
Cardiac arrest (Cardiac disorders) | 4 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 4 | 3 | 8
Coronary artery disease (Cardiac disorders) | 2 | 1 | 2
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 2 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 3 | 0
Blindness transient (Eye disorders) | 0 | 2 | 2
Choroidal neovascularisation (Eye disorders) | 1 | 1 | 2
Dry age-related macular degeneration (Eye disorders) | 0 | 3 | 3
Glaucoma (Eye disorders) | 1 | 0 | 1
Neovascular age-related macular degeneration (Eye disorders) | 2 | 1 | 4
Open angle glaucoma (Eye disorders) | 0 | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0
Uveitic glaucoma (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 10 | 13 | 18
Visual impairment (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 2 | 0
Complication associated with device (General disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 3 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 1
Endometritis (Infections and infestations) | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 4 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 2
Kidney infection (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 3 | 5
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Urosepsis (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 4 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incomplete spinal fusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 3 | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
International normalised ratio abnormal (Investigations) | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 10 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Laryngeal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 1
Coma (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 6 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2
Bladder cyst (Renal and urinary disorders) | 1 | 0 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Fracture treatment (Surgical and medical procedures) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 2 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 1 | 1
Posterior capsule opacification (Eye disorders) | 1 | 0 | 0
Visual acuity reduced transiently (Eye disorders) | 0 | 2 | 1
Hypertension (Vascular disorders) | 0 | 1 | 2
Stent-graft endoleak (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 2
Device malfunction (Product Issues) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Comparator (N=318) | Lampalizumab Q4W (N=329) | Lampalizumab Q6W (N=323)
Conjunctival haemorrhage (Eye disorders) | 84 | 112 | 97
Eye pain (Eye disorders) | 30 | 55 | 36
Vitreous detachment (Eye disorders) | 24 | 37 | 31
Cataract (Eye disorders) | 25 | 23 | 25
Retinal haemorrhage (Eye disorders) | 14 | 24 | 22
Dry eye (Eye disorders) | 16 | 19 | 16
Vitreous floaters (Eye disorders) | 5 | 29 | 26
Blepharitis (Eye disorders) | 11 | 26 | 15
Vision blurred (Eye disorders) | 15 | 18 | 12
Posterior capsule opacification (Eye disorders) | 11 | 20 | 11
Diarrhoea (Gastrointestinal disorders) | 5 | 18 | 8
Nasopharyngitis (Infections and infestations) | 46 | 45 | 36
Urinary tract infection (Infections and infestations) | 22 | 33 | 14
Bronchitis (Infections and infestations) | 16 | 25 | 32
Upper respiratory tract infection (Infections and infestations) | 20 | 19 | 13
Influenza (Infections and infestations) | 13 | 23 | 14
Fall (Injury, poisoning and procedural complications) | 41 | 47 | 28
Intraocular pressure increased (Investigations) | 7 | 50 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 22 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 18 | 14
Headache (Nervous system disorders) | 11 | 20 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 26 | 10
Hypertension (Vascular disorders) | 26 | 27 | 22

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor because the compound had demonstrated lack of efficacy. Thus, not all participants in this study completed the full duration of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-09-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT02247531/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT02247531/SAP_001.pdf